CLINICAL TRIAL: NCT06217679
Title: Comparing the Effects of Different Types of Exercise on Glucose Handling and Muscle Metabolism in Young Males and Females
Brief Title: Comparing the Effects of Different Types of Exercise on Glucose Handling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ORE #22477
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Glycemic Control; Insulin Sensitivity; Sex Differences
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Oral Glucose Tolerance Test (Experimental): This visit will include a baseline OGTT to be used as a pre-exercise baseline measure for each of the arms. Participants will then consume a 75g glucose beverage (Trutol, Thermo Scientific) and blood samples will be drawn at 0, 10, 20, 30, 45, 60, 75, 90 and 120 minutes post consumption.
  Interventions: Other: Control Oral Glucose Tolerance Test; Other: Mixed Exercise
- High intensity interval exercise (HIIE) (Experimental): Participants performed a High intensity interval exercise (HIIE) bout which includes 10 x 1 min at 90% maximum heart rate (HRmax) with 5 min warm up and 5 min cool down at 50watts (low state steady cycling). 90mins following the exercise bout participants will undergo another oral glucose tolerance test.
  Interventions: Other: Control Oral Glucose Tolerance Test; Other: Mixed Exercise
- Moderate intensity continuous exercise (MICE) (Experimental): Participants performed a Moderate intensity continuous exercise (MICE) bout which includes 30 min at 65% maximal aerobic capacity (VO2max). 90mins following the exercise bout participants will undergo another oral glucose tolerance test.
  Interventions: Other: Control Oral Glucose Tolerance Test; Other: Mixed Exercise
- Low-load, high-repetition resistance exercise (LL-HR) (Experimental): Participants performed a Low-load, high-rep resistance exercise (LL-HR) bout which includes a whole body resistance exercise bout, 3 sets at 30% maximum strength (1RM) for leg press, knee extension, hamstring curl, lat pulldown, shoulder press, chest press, 20-25 reps, last set to failure. 90mins following the exercise bout participants will undergo another oral glucose tolerance test.
  Interventions: Other: Control Oral Glucose Tolerance Test; Other: Mixed Exercise

INTERVENTIONS:
Other: Control Oral Glucose Tolerance Test — control oral glucose tolerance test
Other: Mixed Exercise — exercise performed in randomized order

SUMMARY:
The purpose of the proposed study is to compare the acute effects of different types of exercise modalities on glucose handling in young, healthy males and females. The exercise modalities that will be compared include: a high intensity interval exercise (HIIE) protocol, a moderate intensity continuous exercise (MICE) protocol and a low-load, high-repetition (LL-HR) resistance exercise protocol.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of different exercise modalities (High intensity interval exercise, Moderate intensity continuous exercise, and Low-load-high repetition resistance exercise) on blood sugar control in young healthy, males and females. To test this theory, a sugar challenge (oral glucose tolerance test - OGTT) will be performed during the pre-testing visit to determine the baseline blood sugar response. An OGTT will also be performed 2 hours after each single exercise session to determine how each type of exercise affects the blood sugar response. Investigators will take multiple blood samples throughout the trial to allow us to measure blood sugar, insulin and concentrations and oxidative stress. Muscle biopsies will be taken before and after each exercise bout so that investigators can examine the underlying mechanisms that contribute to the effectiveness of the different types of exercise on blood sugar control. Investigators will also use an ultrasound to measure factors related to of cardiovascular health such as artery stress and vascular conductance during the exercise bouts. Direct benefits of this study include characterizing sex differences of blood sugar handling after single exercise sessions. This study could have direct benefits on deterring the effectiveness of different forms of exercise on blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

* In order to participate in this study, participants must be a healthy man or woman between the ages of 18 and 30 years.

Exclusion Criteria:

* Presence of chronic health condition(s) [i.e. metabolic (i.e. Type 1 or type 2 diabetes), cardiovascular (i.e hypertension), respiratory (i.e. chronic pulmonary obstructive disorder) or digestive (i.e. ulcerative colitis) disorders.

  * Are pregnant, or suspect that they may be pregnant, or nursing
  * Inability to complete the single exercise sessions.
  * Regularly participate in cardiovascular (>3 sessions/week) or resistance training (>2 sessions/week) exercise.
  * Have an allergy to local anesthetic (or family history of allergy)
  * Have undergone a barium swallow or an infusion of a contrast agent in the past 3 weeks
  * Are taking prescription anti-coagulant or anti-platelet medications (e.g., warfarin, heparin, clopidogrel)
  * Inability to exercise as suggested by the get active questionnaire (GAQ)
  * BMI > 27 kg/m2

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Blood insulin change | 120mins
  To assess the effect of sex and exercise on basal and post-exercise blood insulin
Blood glucose change | 120mins
  To assess the effect of sex and exercise on basal and post-exercise blood glucose.
Blood c-peptide change | 120mins
  To assess the effect of sex and exercise on basal and post-exercise blood c-peptide.
Insulin sensitivity change | 120mins
  Assess the changes in insulin sensitivity pre to post exercise

SECONDARY OUTCOMES:
TBC1 domain family member 4 change (TBC1D4) | 35mins
  examine protein content changes from pre to post exercise
TBC1 domain family member 1 change (TBC1D1) | 35mins
  examine protein content changes from pre to post exercise
protein kinase B change | 35mins
  examine protein content changes from pre to post exercise
5' adenosine monophosphate-activated protein kinase change | 35mins
  examine protein content changes from pre to post exercise
glucose transporter 4 change (GLUT4) | 35mins
  examine protein content changes from pre to post exercise
estrogen concentration | 30mins
  to assess the differences in estrogen concentration between males and females
progesterone concentration | 30mins
  to assess the differences in progesterone concentration between males and females

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Beaudry KM, Surdi JC, Pancevski K, Tremblay C, Devries MC. Greater glycemic control following low-load, high-repetition resistance exercise compared with moderate-intensity continuous exercise in males and females: a randomized control trial. Appl Physiol Nutr Metab. 2024 Jul 1;49(7):943-955. doi: 10.1139/apnm-2023-0353. Epub 2024 Mar 22. PMID 38518263